CLINICAL TRIAL: NCT04031664
Title: A Clinical Study on Qianjin Capsule of Gynaecology Combined With Antibiotics for Pelvic Inflammatory Diseases (Damp-heat Stasis and Qi Deficiency Syndrome)：a Randomized, Double Blind, Parallel Control of Positive Drugs, Multi-center Clinical Study
Brief Title: A Clinical Study on Qianjin Capsule of Gynaecology Combined With Antibiotics for Pelvic Inflammatory Diseases (Damp-heat Stasis and Qi Deficiency Syndrome)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); Peking University First Hospital (Other); Beijing Obstetrics and Gynecology Hospital (Other); Longhua Hospital (Other); Third Hospital of Peking University (Unknown); Peking Union Medical College Hospital (Other); First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine (Unknown); Shenzhen Maternal and Child Health Hospital (Unknown); First Affiliated Hospital of Heilongjiang Chinese Medicine University (Other); Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy director, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Qianjin Capsule
Record Dates: First submitted 2019-07-11; First posted 2019-07-24 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Pelvic Inflammatory Diseases
Keywords: Qianjin Capsule of Gynaecology; efficacy and safety; recurrence rate; randomized; double blind; parallel control; multi-center clinical study
MeSH Terms: conditions — Pelvic Inflammatory Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qianjin Capsule of Gynaecology (Experimental): On the basis of the antibiotic levofloxacin + metronidazole for 14 days, Gynecological Qianjin Capsule for 28 days.
  One of the levofloxacin quinolones has broadspectrum antimicrobial activity and strong antimicrobial activity. Metronidazole is mainly used to treat or prevent systemic or local infections caused by the abovementioned anaerobes, such as anaerobic infections in abdominal cavity, digestive tract, female reproductive system, lower respiratory tract, skin and soft tissue, bone and joint, etc.
  Interventions: Drug: Qianjin Capsule of Gynaecology
- Antibiotics alone group (Placebo Comparator): Levofloxacin + metronidazole for 14 days, and gynecological Qianjin capsule simulator for 28 days.
  One of the levofloxacin quinolones has broadspectrum antimicrobial activity and strong antimicrobial activity. It has strong antimicrobial activity against most Enterobacteriaceae bacteria, such as Escherichia coli, Klebsiella, Proteus, Salmonella, Shigella and Haemophilus influenzae, Legionella pneumophila, Neisseria gonorrhoeae and other gramnegative bacteria. Bacterial activity. Metronidazole is mainly used to treat or prevent systemic or local infections caused by the abovementioned anaerobes, such as anaerobic infections in abdominal cavity, digestive tract, female reproductive system, lower respiratory tract, skin and soft tissue, bone and joint, etc.
  Interventions: Drug: Qianjin Capsule of Gynaecology

INTERVENTIONS:
Drug: Qianjin Capsule of Gynaecology — To evaluate the short-term and long-term efficacy of traditional Chinese medicine of Qianjin Capsule of Gynaecology in reducing the use of antibiotics, reducing the risk of clinical use of drugs.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety of Qianjin Capsule of Gynaecology combined with antibiotics for pelvic inflammatory diseases (Damp-heat Stasis and Qi Deficiency Syndrome) for the short-term and long-term efficacy of traditional Chinese medicine in reducing the use of antibiotics, reducing the risk of clinical use of drugs.

ELIGIBILITY:
Inclusion Criteria:

* (1) Women aged 20-50;
* (2) Sexual History ;
* (3) According to the diagnostic criteria of pelvic inflammatory diseases: according to the Diagnosis and Treatment Criteria of Pelvic Inflammatory Diseases (2014), the following specifications are as follows: A. uterine tenderness, or adnexal tenderness, or cervical lifting pain; B. axillary body temperature < 38 C. blood routine white blood cell count < 1.1 times the upper limit of normal value; D. blood routine neutrophil percentage < 90%; All of the above four items are available. Exclusion Criteria:
* (4)4<McCormack<12;
* (5)TCM syndrome differentiation for damp-heat stagnation and Qi deficiency syndrome, A. lower abdominal pain; B. excessive amount of belt, yellow color, or odor; C. fatigue; D. tongue red, greasy fur, or with teeth marks, or blood stasis spots; the above four items are all available;
* (6)Those who agree to participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

* (1) Pregnant or recent (within 6 months) pregnant women, lactating women ;
* (2) To identify the pathogen as Neisseria gonorrhoeae;
* (3) Symptoms related to appendicitis, ectopic pregnancy, torsion or rupture of ovarian cyst pedicle, gastroenteritis, endometriosis, adenomyosis, trichomonal vaginitis, vulvovaginal candidiasis, bacterial vaginosis, etc.;
* (4)Those with critical condition or surgical indications, such as fallopian tube and ovary abscess, pelvic abscess, diffuse peritonitis, septicemia;
* (5)In patients with severe primary diseases such as heart, brain and hematopoietic system, ALT of liver function is higher than the upper limit of normal value, and Cr of renal function is higher than the upper limit of normal value;
* (6)One month before admission, Chinese and Western medicines were used to treat the disease, which made it difficult to judge the efficacy of drugs;
* (7)Anaphylactic constitution or persons known to be allergic to the medicines and their components used in this test ;
* (8)Researchers do not consider it appropriate to participate in this clinical trial;
* (9)Suspected or true history of alcohol and drug abuse, or other pathological changes or conditions that reduce the likelihood of enrollment or complicate enrollment, such as frequent changes in the working environment, unstable living environment, etc., are liable to lead to lost interviews, according to the judgement of researchers;
* (10)Participation in other clinical researchers within 3 months before admission;
* (11)Patients with suspected or confirmed quinolone contraindications, central or peripheral neuropathy, epilepsy, and depression

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Estimated)
Dates: Start 2019-08-02 (Estimated); Primary Completion 2019-08-02 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The MCCormack scale scores of 184 subjects will be assessed | Change from base line on the 56 days after discontinuation
  assessment of the 70% reduction rate after treatment

SECONDARY OUTCOMES:
The neutrophils of 184 participants will be assessed | Change from base line on the 28 days of medication and 56 days after discontinuation
  assessment of neutrophils returning to normal reference range
The whole blood reduced viscosity from hemorheological tests of 184 participants will be assessed | Change from base line on the 28 day of medication.
  assessment of whole blood viscosity returning to normal reference range
The plasma viscosity from hemorheological tests of 184 participants will be assessed | Change from base line on the 28 day of medication.
  assessment of the plasma viscosity returning to normal reference range
The fibrinogen determination from hemorheological tests of 184 participants will be assessed | Change from base line on the 28 day of medication.
  assessment of the fibrinogen determination returning to normal reference range
The CRP of 184 participants will be assessed | Change from base line on the 28 day of medication.
  assessment of the CRP returning to normal reference range
The volume of liquid on B-mode of 184 subjects will be assessed | After 28 days of medication
  The changes of the volume of liquid on B-mode at different observation points before and after treatment will be assessed
The white blood cells of 184 participants will be assessed | Change from base line on the 28 days of medication and 56 days after discontinuation
  assessment of the white blood returning to normal reference range
The TCM syndrome scores of 184 subjects will be assessed | Change from base line on the 56 days after discontinuation
  assessment of the 70% reduction rate after treatment
The VAS score of 184 subjects will be assessed | Change from base line on the 56 days after discontinuation
  assessment of the 70% reduction rate after treatment

OTHER OUTCOMES:
Adverse events | Change from base line on the 21 day of medication and from 28 days on 56 days after the end of
  Observe the incidence of adverse events after medication
Change of liver function | Change from base line on the 21 day of medication and from 28 days on 56 days after the end of
  To observe whether ALT and AST are within the normal reference range after medication.
Change of renal function | Change from base line on the 21 day of medication and from 28 days on 56 days after the end of
  To observe whether creatinine and urea nitrogen are within the normal reference range after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yanming Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese

IPD SHARING:
Plan to Share IPD: No